CLINICAL TRIAL: NCT06285136
Title: The Second Affiliated Hospital of Kunming Medical University
Brief Title: Safety and Efficacy of Venetoclax Combination With Decitabine(DEC3-VEN) in the Treatment of AML in the Adult
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other); Handan Central Hospital (Other); Taian City Central Hospital (Other); Tianjin People's Hospital (Other); Guizhou Provincial People's Hospital (Other); Central South University (Other); Western Theater General Hospital (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); Chengdu Jingdongfang Hospital (Unknown)
Responsible Party: Principal Investigator, ZePing Zhou, Director, The Second Affiliated Hospital of Kunming Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEN-PJ-KE-2024-15
Record Dates: First submitted 2024-02-18; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Acute Myeloid Leukemia, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax in combination with Decitabine (+-sorafenib) (Experimental): Venetoclax in combination with decitabine (+-sorafenib) Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-14 Decitabine (DEC) 20mg/m2/q8h, d4-6 (infusion time >2h) Sorafenib 800mg/d, d8-14 (only for FLT3/ITD mutation positive patients)
  Interventions: Procedure: DEC3-VEN

INTERVENTIONS:
Procedure: DEC3-VEN — Venetoclax in combination with decitabine (+-sorafenib) Venetoclax (VEN) 100mg d1, 200mg d2, 400mg d3-14 Decitabine (DEC) 20mg/m2/q8h, d4-6 (infusion time >2h) Sorafenib 800mg/d, d8-14 (only for FLT3/ITD mutation positive patients)

SUMMARY:
This study proposes to conduct a prospective, multicenter, single-arm study to explore the efficacy and safety of venetoclax in combination with high-dose decitabine (DEC3-VEN) in new diagnosed adult patients with AML, and to provide evidence for the optimal selection of clinical treatment regimens, which is planned to be conducted in 10 research centers across the country.

ELIGIBILITY:
Inclusion Criteria:

Subjects suitable for enrollment in this study must meet all of the following criteria:

1. meet the World Health Organization diagnostic criteria (WHO2022 criteria) other than APL or carrying one of the abnormal karyotypes such as t(8;21)/(RUNX1::RUNX1TI), inv(16)(p13.1q22), t(16;16) (p13.1q22), t(16;16)/CBFβ::myh11), etc. Patients with acute myeloid leukemia other than those with one of the abnormal karyotypes such as t(16;16)/CBFβ::myh11
2. Patients with AML not otherwise classified under the World Health Organization AML classification, except for acute myeloproliferative disorder with myelofibrosis and myeloid sarcoma;
3. patients of either sex, age greater than or equal to 16 years and less than 65 years, with a primary diagnosis of AML, who are considered suitable for intensive chemotherapy;
4. Eastern Cooperative Oncology Group (ECOG) physical status ≤ 2 at enrollment;
5. the patient has not received prior treatment for AML (except hydroxyurea and Ara-C <1.0 g/d for tumor composite reduction);
6. passes the following laboratory test markers (performed within 7 days prior to treatment):1) aspartate aminotransferase (ALT), alanine aminotransferase (AST), and alkaline phosphatase (ALP) ≤ 3 x upper limit of normal (ULN), serum bilirubin ≤ 2 x ULN; and serum cardiac enzymes < 2.0 x ULN; unless leukemic organ involvement is considered.2) Creatinine ≥ 30 mL/min, calculated by the Cockcroft Gault formula or measured by 24-hour urine collection
7. Female subjects of childbearing potential must have a negative pregnancy test result within 72 hours prior to the start of treatment; no pregnancy is planned during the study and within 6 months of the last dose of study drug, and a negative urine or serum pregnancy test result at screening. Men must use latex condoms during any sexual contact with WOCBP, even if they have undergone a successful vasectomy, and must agree to avoid childbearing (during treatment and within 6 months of the last dose of study drug);
8. have a life expectancy of more than 2 months;
9. informed consent must be signed prior to the start of all specific study procedures, either by the patient himself/herself or by a member of his/her immediate family; if, in view of the patient's medical condition, his/her own signature would not be conducive to the treatment of his/her medical condition, the informed consent will be signed by his/her legal guardian or by a member of the patient's immediate family.

Exclusion Criteria:

Subjects may not be enrolled in this study if they meet any of the following criteria:

1. AML with BCR-ABL1; or CML acute stage;
2. Treatment-naïve patients (is defined as having received prior induction chemotherapy regardless of efficacy);
3. Subjects with acute total myelopathy with myelofibrosis or myeloid sarcoma as defined by WHO 2016;
4. Secondary leukemia (primarily those whose World Health Organization (WHO 2016) AML classification falls into the subcategory of treatment-related AML and those with a history of prior MDS and/or MPD);
5. concurrent other hematologic diseases (e.g., hemophilia, myelofibrosis, etc., who are considered unsuitable for enrollment by the investigator; those who have previous blood abnormalities but have ever had bone marrow tests except for MDS and MPD are allowed to be enrolled);
6. Pregnant or lactating patients;
7. Those who are allergic to any drugs involved in this study;
8. Have used strong or moderate CYP7A inducers within 3 days prior to the start of study treatment;
9. concurrent malignant tumors of other organs (those requiring treatment);
10. Significantly abnormal hepatic or renal function beyond the enrollment criteria;
11. Active heart disease, defined as one or more of the following:1) Myocardial infarction less than 6 months from study entry; 2) A history of arrhythmia requiring medication or severe clinical symptoms; 3) Uncontrolled or symptomatic congestive heart failure (> NYHA class 2); 4) Uncontrolled or symptomatic angina;5) Left ventricular ejection fraction below the lower limit of the normal range;
12. severe infectious diseases (untreated tuberculosis, pulmonary aspergillosis), patients with known infection with human immunodeficiency virus (HIV) or active hepatitis B or C; subjects with uncontrolled treatment.
13. Subjects with evidence of central nervous system leukemia prior to treatment;
14. Subjects with epilepsy requiring medication, dementia, or other abnormal mental states that are unable to understand or follow the regimen;
15. Conditions that limit oral drug intake or gastrointestinal absorption;
16. those who, in the opinion of the investigator, are not suitable for enrollment;

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
ORR | up to 24 months
  ORR (include CR, CRi, MLFS, PR) of the first course of Venetoclax in combination with high-dose decitabine for the treatment of newly-diagnosed AML adult patients.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 24 months
  defined as the time period from initiation of study medication to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Kunming Medical University., Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Del Poeta G, Venditti A, Del Principe MI, Maurillo L, Buccisano F, Tamburini A, Cox MC, Franchi A, Bruno A, Mazzone C, Panetta P, Suppo G, Masi M, Amadori S. Amount of spontaneous apoptosis detected by Bax/Bcl-2 ratio predicts outcome in acute myeloid leukemia (AML). Blood. 2003 Mar 15;101(6):2125-31. doi: 10.1182/blood-2002-06-1714. Epub 2002 Nov 7. PMID 12424199
- [Background] Mei M, Aldoss I, Marcucci G, Pullarkat V. Hypomethylating agents in combination with venetoclax for acute myeloid leukemia: Update on clinical trial data and practical considerations for use. Am J Hematol. 2019 Mar;94(3):358-362. doi: 10.1002/ajh.25369. Epub 2018 Dec 13. PMID 30499168
- [Background] Pettit K, Odenike O. Defining and Treating Older Adults with Acute Myeloid Leukemia Who Are Ineligible for Intensive Therapies. Front Oncol. 2015 Dec 14;5:280. doi: 10.3389/fonc.2015.00280. eCollection 2015. PMID 26697412
- [Background] Wei AH, Strickland SA Jr, Hou JZ, Fiedler W, Lin TL, Walter RB, Enjeti A, Tiong IS, Savona M, Lee S, Chyla B, Popovic R, Salem AH, Agarwal S, Xu T, Fakouhi KM, Humerickhouse R, Hong WJ, Hayslip J, Roboz GJ. Venetoclax Combined With Low-Dose Cytarabine for Previously Untreated Patients With Acute Myeloid Leukemia: Results From a Phase Ib/II Study. J Clin Oncol. 2019 May 20;37(15):1277-1284. doi: 10.1200/JCO.18.01600. Epub 2019 Mar 20. PMID 30892988
- [Background] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659